CLINICAL TRIAL: NCT07065162
Title: Combined Effects of Subtle Touch Technique and Active Cycle of Breathing Technique in COPD
Brief Title: Effects of Subtle Touch Technique and Active Cycle of Breathing Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0354
Record Dates: First submitted 2025-06-11; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subtle Touch Technique with Active Cycle of Breathing Technique (Experimental): Group A will receive 3 cycles of ACBT along with subtle touch technique for 15 minutes 3 times daily for 8 weeks, in addition to the standard COPD care and medication.
  Interventions: Other: Subtle Touch Technique
- Active Cycle of Breathing Technique (Active Comparator): Group B will receive 3 cycles of ACBTs technique for 15 minutes 3 times daily for 8 weeks, along with standard COPD care and medication.
  Interventions: Other: Active Cycle of Breathing Technique

INTERVENTIONS:
Other: Subtle Touch Technique — 3 cycles of ACBT along with subtle touch technique for 15 minutes 3 times daily for 8 weeks, in addition to the standard COPD care and medication.
  Other Names: Active Cycle of Breathing Technique
  Arms: Subtle Touch Technique with Active Cycle of Breathing Technique
Other: Active Cycle of Breathing Technique — 3 cycles of ACBTs technique for 15 minutes 3 times daily for 8 weeks, along with standard COPD care and medication.
  Arms: Active Cycle of Breathing Technique

SUMMARY:
COPD is a disease state characterized by the presence of airflow obstruction due to chronic bronchitis or emphysema. Subtle Touch, also known as Calatonia, involves a profound relaxation approach that regulates muscle tension and fosters physical and psychological equilibrium in patients. The study will employ a randomized controlled trial, with total 40 participants divided into two groups. Group A will receive ACBTs three times daily for fifteen minutes for eight weeks. Group B will receive ACBT along with subtle touch technique for three times daily for fifteen minutes for eight weeks. The nonprobability convenient sampling technique, followed by random allocation using sealed opaque enveloped method.The inclusion criteria will be focusing on patients of 45 to 60 years of age, patients with mild to moderate COPD (according to Gold Criteria) and both male and female. While exclusion criterion includes musculoskeletal disorders, any recent chest injuries, lung infections and pulmonary hypertension. The methodology will involve 8-week intervention period, conducted at pulmonology department of Jinnah hospital, with participants in each group receiving instruction and support in their respective breathing techniques. All patients will be assessed using Digital Spirometer (to evaluate pulmonary functions), Breathlessness Cough and Sputum Scale BCSS (to evaluate sputum diary of patients), Modified Borg Dyspnea Scale and St. George's Respiratory Questionnaire (SGRQ). The data analysis will be done by using SPSS version 25. After assessing Combined Effects of ACBT and Subtle Touch Technique in COPD normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

DETAILED DESCRIPTION:
COPD is a disease state characterized by the presence of airflow obstruction due to chronic bronchitis or emphysema. In 2018, approximately 5.1% of adults (equivalent to around 12.8 million individuals) received a COPD diagnosis. Subtle Touch, also known as Calatonia, involves a profound relaxation approach that regulates muscle tension and fosters physical and psychological equilibrium in patients. It entails gentle stimulation of nerve receptor-rich areas of the body, promoting muscle relaxation and potentially improving respiratory muscle function. The study will employ a randomized controlled trial, with total 40 participants divided into two groups. Group A will receive ACBTs three times daily for fifteen minutes for eight weeks.

Group B will receive ACBT along with subtle touch technique for three times daily for fifteen minutes for eight weeks. The nonprobability convenient sampling technique, followed by random allocation using sealed opaque enveloped method, ensures a diverse yet unbiased sample. The inclusion criteria will be focusing on patients of 45 to 60 years of age, patients with mild to moderate COPD (according to Gold Criteria) and both male and female. While exclusion criterion includes musculoskeletal disorders, any recent chest injuries, lung infections and pulmonary hypertension. The methodology will involve 8-week intervention period, conducted at pulmonology department of Jinnah hospital, with participants in each group receiving instruction and support in their respective breathing techniques. All patients will be assessed using Digital Spirometer (to evaluate pulmonary functions), Breathlessness Cough and Sputum Scale BCSS (to evaluate sputum diary of patients), Modified Borg Dyspnea Scale and St. George's Respiratory Questionnaire (SGRQ). The data analysis will be done by using SPSS version 25. After assessing

1 Combined Effects of ACBT and Subtle Touch Technique in COPD normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 to 65
* Patients with mild to moderate COPD (according to Gold Criteria)
* Both male and female (18).

Exclusion Criteria:

* Musculoskeletal disorders
* Any recent chest injuries
* Lung infections
* Pulmonary hypertension (18)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
St. George's Respiratory Questionnaire (SGRQ) | 8 weeks
  Patients were assessed through the help of Saint George respiratory Questionnaire (SGRQ) which is disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scaling includes Part
  1: (Symptoms) frequency & severity with 1, 3 or 12-month recall (best performance with 3- and 12-month recall) Part 2: (Activity and Impacts) Activities that cause or are limited by breathlessness; Impact components (social functioning, psychological disturbances resulting from airways disease) refer to current state as the recall. Validity include significant correlations between total score and presence of cough, sputum, and wheeze
Breathlessness, Cough and Sputum Scale (BCSS) | 8 weeks
  The Sputum Diary will be assessed using the Breathlessness, Cough and Sputum Scale (BCSS). This scale consists of three items that patients report on: breathlessness, cough, and sputum. Participants rate each symptom on a 5-point Likert scale ranging from 0 to 4, where higher scores indicate more severe symptoms. The total score ranges from 0 to 12 The scale has been validated for its reliability and validity, and its suitability for measuring the errors associated with BCSS has been examined. Internal consistency and reproducibility (test-retest reliability) were assessed using Cronbach's alpha coefficient. Discriminant validity was tested using two methods: analysis of variance (ANOVA) with post Hoc Scheffé test to determine variations in BCSS scores based on disease severity levels
Modified Borg Dyspnea Scale | 8 weeks
  Modified Borg Dyspnea scale, a reliable and valid tool, will be used to report the intensity of Dyspnea related symptoms experienced by patients. Modified Borg Scale: 11-point scale ranges from 0 (no dyspnea to 10 (max dyspnea). It has been found it has been shown to be reliable for quantifying dyspnea in trial patients

SECONDARY OUTCOMES:
Digital Spirometer | 8 weeks
  Spirometry is a physiological test that measures the ability to inhale and exhale air relative to time. Spirometry is a diagnostic test of several common respiratory disperses such as asthma and chronic obstructive pulmonary disease (COPD).

CONTACTS AND LOCATIONS:
Overall Officials: iram nawaz, mphill, Principal Investigator — Riphah International University
Locations (1):
- Gulab Devi Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang W, Li F, Li C, Meng J, Wang Y. Focus on Early COPD: Definition and Early Lung Development. Int J Chron Obstruct Pulmon Dis. 2021 Nov 25;16:3217-3228. doi: 10.2147/COPD.S338359. eCollection 2021. PMID 34858022
- [Background] Melam GR, Zakaria A, Buragadda S, Sharma D, Alghamdi MA. Comparison of Autogenic Drainage & Active Cycle Breathing Techniques on FEV1, FVC & PERF in Chronic Obstructive Pulmonary Disease. World Applied Sciences Journal. 2012;20(6):818-22.
- [Background] Lewis LK, Williams MT, Olds TS. The active cycle of breathing technique: a systematic review and meta-analysis. Respir Med. 2012 Feb;106(2):155-72. doi: 10.1016/j.rmed.2011.10.014. Epub 2011 Nov 18. PMID 22100537
- [Background] Sandelowsky H, Weinreich UM, Aarli BB, Sundh J, Hoines K, Stratelis G, Lokke A, Janson C, Jensen C, Larsson K. COPD - do the right thing. BMC Fam Pract. 2021 Dec 11;22(1):244. doi: 10.1186/s12875-021-01583-w. PMID 34895164
- [Background] Cai S, Yao J, Han M, Luo X, Yu Y, Lu X, Xiang X, Huang L. The effect of cognition in combination with an ACBT on dyspnea-related kinesiophobia in patients with moderate to severe COPD: Quasirandomized controlled trial study. Geriatr Nurs. 2024 Mar-Apr;56:138-147. doi: 10.1016/j.gerinurse.2024.01.002. Epub 2024 Feb 10. PMID 38342002